CLINICAL TRIAL: NCT06776107
Title: Factors Associated With Mortality in Brain Injury at the Intensive Care Unit. A Cross-sectional Trial, 2019-2023 (TraVi II)
Brief Title: Mortality in Brain Injury at the Intensive Care Unit (TraVi II)
Acronym: TraVi_II
Status: Completed | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, ICU chief of staff, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2024_01_TCE
Record Dates: First submitted 2024-12-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Traumatic Brain Injuries
Keywords: Brain Injuries; Traumatic Brain Injuries; Brain Concussion; Traffic Accidents; Critical Care; Colombia
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Brain Concussion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mortality: Survival
  Interventions: Other: Risk factor present

INTERVENTIONS:
Other: Risk factor present — Demographic, and severity.

SUMMARY:
Introduction: traumatic brain injuries are a leading cause of disability and mortality in the young population, associated mainly with traffic road accidents and violent wounds. The study aimed to analyze factors related to the mortality in patients with brain injury admitted to the intensive care unit.

Methodology: Between 2019 and 2024, an analytical cross-sectional trial at Hospital Departamental de Villavicencio, Colombia was performed. Information was selected from the intensive care unit (ICU) database. Variables of interest and outcomes, such as mortality and ICU length of stay, were identified. The comparison was performed with the software Prism® for Mac iOS and Wizard® for the predictive model.

Results: The study will show the factors associated with mortality of brain injury patients admitted to the intensive care unit.

DETAILED DESCRIPTION:
Objective: The study aimed to analyze factors related to the mortality in patients with brain injury admitted to the intensive care unit.

Methodology: Between 2019 and 2024, an analytical cross-sectional trial at Hospital Departamental de Villavicencio, Colombia, a reference center for the Colombian Orinoco region with 400 hospital beds and 53 polyvalent ICU beds was performed. Information was selected from 2,154 admission registers in the intensive care unit (ICU) database. Data of admissions considered for review were from patients with diagnostic codes of brain injury, brain edema, polytrauma, ventilatory failure, neurogenic shock, and traumatic subarachnoid hemorrhage. All the registries with codes S00-S09 from the 10th revision of the International Diseases Classification from the World Health Organization were reviewed. Variables of interest and outcomes, such as mortality and ICU length of stay, were identified. The comparison was performed with the software Prism® for Mac iOS and Wizard® for the predictive model.

Results: The study will show the factors associated with mortality of brain injury patients admitted to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury.
* Admitted to the intensive care unit.

Exclusion Criteria:

* Remission from another hospital.
* Decease for causes other than the brain injury.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was patients with traumatic brain injury who were admitted to the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
ICU mortality | 30 days
  Mortality at the ICU

SECONDARY OUTCOMES:
ICU length of stay | 30 days
  Length of stay at the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Principal Investigator — Hospital Departamental de Villavicencio
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: No
It contains sensible information about patients.

REFERENCES:
- [Result] Ortega Zufiria JM, Prieto NL, Cuba BC, Degenhardt MT, Nunez PP, Lopez Serrano MR, Lopez Raigada AB. [Mild head injury]. Surg Neurol Int. 2018 Jan 22;9(Suppl 1):S16-S28. doi: 10.4103/sni.sni_371_17. eCollection 2018. Spanish. PMID 29430327
- [Result] Gonzalez-Robledo J, Martin-Gonzalez F, Moreno-Garcia M, Sanchez-Barba M, Sanchez-Hernandez F. Prognostic factors associated with mortality in patients with severe trauma: from prehospital care to the Intensive Care Unit. Med Intensiva. 2015 Oct;39(7):412-21. doi: 10.1016/j.medin.2014.06.004. Epub 2014 Sep 2. English, Spanish. PMID 25189470
- [Result] Fonseca J, Liu X, Oliveira HP, Pereira T. Mortality prediction using medical time series on TBI patients. Comput Methods Programs Biomed. 2023 Dec;242:107806. doi: 10.1016/j.cmpb.2023.107806. Epub 2023 Sep 21. PMID 37832428
- [Result] Buh FC, Sumbele IUN, Maas AIR, Motah M, Pattisapu JV, Youm E, Meh BK, Kobeissy FH, Wang KW, Hutchinson PJA, Taiwe GS. Traumatic Brain Injury in Cameroon: A Prospective Observational Study in a Level I Trauma Centre. Medicina (Kaunas). 2023 Aug 28;59(9):1558. doi: 10.3390/medicina59091558. PMID 37763678
- [Result] Domensino AF, Tas J, Donners B, Kooyman J, van der Horst ICC, Haeren R, Aries MJH, van Heugten C. Long-Term Follow-Up of Critically Ill Patients With Traumatic Brain Injury: From Intensive Care Parameters to Patient and Caregiver-Reported Outcome. J Neurotrauma. 2024 Jan;41(1-2):123-134. doi: 10.1089/neu.2022.0474. Epub 2023 Oct 10. PMID 37265152
- [Result] Launey Y, Coquet A, Lasocki S, Dahyot-Fizelier C, Huet O, Le Pabic E, Roquilly A, Seguin P. Factors associated with an unfavourable outcome in elderly intensive care traumatic brain injury patients. a retrospective multicentre study. BMC Geriatr. 2022 Dec 30;22(1):1004. doi: 10.1186/s12877-022-03651-x. PMID 36585608
- [Result] Rowe M, Brown J, Marsh A, Thompson J. Predicting Mortality Following Traumatic Brain Injury or Subarachnoid Hemorrhage: An Analysis of the Validity of Standardized Mortality Ratios Obtained From the APACHE II and ICNARC H-2018 Models. J Neurosurg Anesthesiol. 2023 Jul 1;35(3):292-298. doi: 10.1097/ANA.0000000000000831. Epub 2022 Feb 4. PMID 35125410
- [Result] Luostarinen T, Vehvilainen J, Lindfors M, Reinikainen M, Bendel S, Laitio R, Hoppu S, Ala-Kokko T, Skrifvars M, Raj R. Trends in mortality after intensive care of patients with traumatic brain injury in Finland from 2003 to 2019: a Finnish Intensive Care Consortium study. Acta Neurochir (Wien). 2022 Jan;164(1):87-96. doi: 10.1007/s00701-021-05034-4. Epub 2021 Nov 2. PMID 34725728
- [Result] Rubiano AM, Griswold DP, Jibaja M, Rabinstein AA, Godoy DA. Management of severe traumatic brain injury in regions with limited resources. Brain Inj. 2021 Sep 19;35(11):1317-1325. doi: 10.1080/02699052.2021.1972149. Epub 2021 Sep 7. PMID 34493135
- [Result] Kokkinou M, Kyprianou TC, Kyriakides E, Constantinidou F. A population study on the epidemiology and outcome of brain injuries in intensive care. NeuroRehabilitation. 2020;47(2):143-152. doi: 10.3233/NRE-203111. PMID 32741786
- [Result] Venkatasubba Rao CP, Suarez JI, Martin RH, Bauza C, Georgiadis A, Calvillo E, Hemphill JC 3rd, Sung G, Oddo M, Taccone FS, LeRoux PD; PRINCE Study Investigators. Global Survey of Outcomes of Neurocritical Care Patients: Analysis of the PRINCE Study Part 2. Neurocrit Care. 2020 Feb;32(1):88-103. doi: 10.1007/s12028-019-00835-z. PMID 31486027
- [Result] Pappacena S, Bailey M, Cabrini L, Landoni G, Udy A, Pilcher DV, Young P, Bellomo R. Early dysglycemia and mortality in traumatic brain injury and subarachnoid hemorrhage. Minerva Anestesiol. 2019 Aug;85(8):830-839. doi: 10.23736/S0375-9393.19.13307-X. Epub 2019 Feb 7. PMID 30735020
- [Result] Volovici V, Ercole A, Citerio G, Stocchetti N, Haitsma IK, Huijben JA, Dirven CMF, van der Jagt M, Steyerberg EW, Nelson D, Cnossen MC, Maas AIR, Polinder S, Menon DK, Lingsma HF. Intensive care admission criteria for traumatic brain injury patients across Europe. J Crit Care. 2019 Feb;49:158-161. doi: 10.1016/j.jcrc.2018.11.002. Epub 2018 Nov 8. PMID 30447560
- [Result] Raj R, Bendel S, Reinikainen M, Hoppu S, Luoto T, Ala-Kokko T, Tetri S, Laitio R, Koivisto T, Rinne J, Kivisaari R, Siironen J, Skrifvars MB. Traumatic brain injury patient volume and mortality in neurosurgical intensive care units: a Finnish nationwide study. Scand J Trauma Resusc Emerg Med. 2016 Nov 8;24(1):133. doi: 10.1186/s13049-016-0320-6. PMID 27821129